CLINICAL TRIAL: NCT02903732
Title: Autism Registry for French Guiana
Acronym: REGUYAUT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier de Cayenne (Other)
Responsible Party: Sponsor
Other Study IDs: REGUYAUT
Record Dates: First submitted 2016-09-06; First posted 2016-09-16 (Estimated); Last update posted 2016-09-16 (Estimated); Status verified 2016-09

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Watchful Waiting

STUDY DESIGN:
Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: observational — registry

SUMMARY:
The objective of the autism registry is to estimate the prevalence of autism in French Guiana in the cohort of children aged 8 years. Secondary objectives are to determine the prevalence of comorbidities, and to determine the theoretical and actual orientation of these children regarding care and education in a territory with significant structural deficits relative to mainland France. The outcomes of this registry will be to guide decision makers in their funding priorities to improve, screening, diagnosis, care and education for children on the autistic spectrum

ELIGIBILITY:
Inclusion Criteria:

* children aged 8 years with a diagnosis of autism spectrum disorder

Exclusion Criteria:

* refusal to participate

Ages: 8 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: children aged 8 years will be the denominator. the numerator is children who are seeking assistance for care or educational purposes at the unique administration dealing with handicap in French Guiana
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2015-09; Primary Completion 2015-09 (Actual); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
autism spectrum disorder | 1 year (the year at age 8)
  the number of 8 year old children with a diagnosis of autism spectrum disorder in a given year relative to the total population of children aged 8 years old in that given year

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier de Cayenne, Cayenne, French Guiana, France